CLINICAL TRIAL: NCT03338088
Title: Evaluation of Adherence to Clinical Treatment of Glaucoma in Patients of a Reference Ophthalmological Hospital in Goiânia
Brief Title: Evaluation of Adherence to Clinical Treatment of Glaucoma
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Instituto de Olhos de Goiania (Other)
Responsible Party: Sponsor
Other Study IDs: INSTITUTO DE OLHOS-MAYRA 2018
Record Dates: First submitted 2017-11-07; First posted 2017-11-09 (Actual); Last update posted 2017-11-21 (Actual); Status verified 2017-11

CONDITIONS: Glaucoma; Drugs
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Evaluation of adherence to clinical treatment of glaucoma in patients of a Reference Ophthalmological Hospital in Goiânia using Morisky Adhesion scale as a validated questionary.

ELIGIBILITY:
Inclusion Criteria: have glaucoma diagnosed -

Exclusion Criteria: not having glaucoma diagnosed

-

Ages: 1 Year to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All pacients that have glaucoma diagnosed that respond the questionary
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2017-11-06 (Actual); Study Completion 2017-12-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of adherence to clinical treatment of glaucoma in patients of a Reference Ophthalmological Hospital in Goiânia | 2 months
  evaluation of the scale

CONTACTS AND LOCATIONS:
Overall Officials: Joao jr Nassaralla, coordinator, Study Director — coordinator
Locations (1):
- Instituto de Olhos de Goiania, Goiânia, Goiás, Brazil

IPD SHARING:
Plan to Share IPD: No